CLINICAL TRIAL: NCT03825250
Title: A Randomised Controlled Trial of Pre-surgery Sodium ValpRoate, for the Prevention of Organ Injury in Cardiac Surgery: THE Val-CARD TRIAL
Brief Title: The Val-CARD Trial
Acronym: Val-CARD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0667; 2018-002076-41 (EudraCT Number); 246126 (Registry Identifier: IRAS); 18/EM/0188 (Other: REC East Midlands)
Record Dates: First submitted 2018-08-31; First posted 2019-01-31 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Valve Disease; Coronary Artery Disease; Organ Failure, Multiple
Keywords: Sodium Valproate; Cardiac Surgery; Organ Injury Prevention
MeSH Terms: conditions — Heart Valve Diseases; Coronary Artery Disease; Multiple Organ Failure | interventions — Valproic Acid

STUDY DESIGN:
Intervention Model Description: Unblinded two phased randomised controlled trial
  * Discovery phase: 4 groups (1 control, 3 treatment)
  * Efficiency phase: 2 groups (1 control, 1 treatment)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Control (No Intervention): Standard of care
- Group B: Sodium Valproate Treatment (Experimental): 15 mg/kg for 1-2 weeks
  Interventions: Drug: Sodium Valproate
- Group C: Sodium Valproate Treatment (Experimental): 15 mg/kg for 4-6 weeks
  Interventions: Drug: Sodium Valproate
- Group D: Sodium Valproate Treatment (Experimental): 25 mg/kg for 4-6 weeks
  Interventions: Drug: Sodium Valproate

INTERVENTIONS:
Drug: Sodium Valproate — Treatment with Sodium Valproate vs. Control Discovery phase - 4 arms: 15 mg/kg for 1-2 weeks; 15mg/kg for 4-6 weeks; 25 mg/kg for 4-6 weeks; Control Efficiency phase - 2 arms: Treatment group selected from previous phase; Control
  Arms: Group B: Sodium Valproate Treatment; Group C: Sodium Valproate Treatment; Group D: Sodium Valproate Treatment

SUMMARY:
The Val-CARD trial aims to answer the question: "Does the drug sodium valproate reduce complications affecting the heart and kidneys in patients having heart operations?" Sodium valproate is a drug commonly used in the treatment of epilepsy. Recently it has been shown to protect against heart and kidney damage in laboratory tests. This has led to trials evaluating whether it can prevent heart and kidney damage in patients. The investigators wish to evaluate whether treatment with sodium valproate for a short period can reduce levels of organ damage following heart surgery by measuring this in blood tests, exercise tests, a special x-ray measuring body fat content, a walk exercise and muscle strength tests. The investigators now want to establish if sodium valproate works by making the heart and kidney more resistant to any injury that results from the use of the heart lung machine.

DETAILED DESCRIPTION:
This trial is a single centre, unblinded, randomised controlled trial of pre-surgery sodium valproate versus standard care (no treatment). The trial has two phases. In the first phase - the dose finding phase, 40 patients will be randomised (1:1:1:1) to three different treatment doses versus a control group of standard care (no treatment). A single sodium valproate dose will be selected based on the evaluation of compliance, toxicity and levels of Histone Deacetylase inhibition. In the second phase, the efficacy of this dose at preventing myocardial and kidney injury will then be compared to untreated controls using a 1:1 randomised parallel group design in a further 82 patients. In an optional research procedure during the efficacy phase of the trial (Phase 2) cardiometabolic status (cardiac function and visceral adiposity) will be evaluated using MRI scanning.

Patients will be screened by the investigators to assess eligibility for entry into the trial. Eligible patients undergoing cardiac surgery with CPB who consent to participate will be randomly allocated using concealed allocation as follows:

In the dose finding phase of the trial patient will be randomised in a 1:1:1:1 ratio to:

1. GROUP A: Standard care (no treatment)
2. GROUP B: Sodium valproate at a target dose of 15 mg/kg per day for 1-2 weeks pre-surgery.
3. Group C: Sodium valproate at a target dose of 15 mg/kg per day for 4-6 weeks pre-surgery.
4. Group D: Sodium valproate at a target dose of 25 mg/kg per day for 4-6 weeks pre-surgery.

In the efficacy phase of the trial patients will be randomised in a 1:1 ratio to:

1. GROUP A: Standard care (no treatment)
2. GROUP B, C or D: Sodium valproate at a target dose as determined by the dose finding phase of the trial.

The Val-CARD Trial proposes to test the overarching hypothesis that pre-surgery administration of sodium valproate will protect patients against organ damage that occurs during cardiac surgery with cardiopulmonary bypass.

The trial will test a number of specific hypotheses:

1. Pre-surgery sodium valproate will reduce the risk of post cardiac surgery organ failure.
2. Short-term (1-2 weeks) pre-surgery treatment with sodium valproate at a target dose of 15mg/kg/day will have different pharmacokinetics but comparable tolerability and protective effects on myocardial and renal signaling to long-term (4-6 weeks) treatment at a target dose of 15mg/kg/ day or 25mg/kg/day.
3. Sodium valproate will reduce the risk of post cardiac surgery myocardial injury by increasing the expression of genes that promote myocardial mitochondrial homeostasis via effects on chromatin histone deacetylation.
4. Sodium valproate will reduce the risk of post cardiac surgery acute kidney injury (AKI) by increasing the expression of genes that promote renal tubular homeostasis.
5. Sodium valproate will reduce the risk of post cardiac surgery endothelial dysfunction by increasing the expression of genes that promote endothelial homeostasis.
6. The trial interventions will be tolerated by patients and will not result in long-term adverse changes in cardiometabolic status.

ELIGIBILITY:
Inclusion Criteria:

* Adult cardiac surgery patients (≥18 years) undergoing cardiac surgery (CABG, Valve, or CABG and Valve) with cardiopulmonary bypass (CPB).
* Able, in the opinion of the investigator, and willing to give informed consent.

Exclusion Criteria:

* Emergency or salvage procedure
* Patients with end stage renal failure defined as an estimated Glomerular Filtration rate (eGFR) <15 mL/min/1.72 m2 calculated from the Modification of Diet in Renal Disease equation,1 or patients who are on long-term haemodialysis or have undergone renal transplantation.
* Patients with persistent or chronic atrial fibrillation.
* Patients with acute liver disease.
* Personal or family history of severe hepatic dysfunction, especially drug related.
* Patients allergic to sodium valproate.
* Patients with thrombocytopaenia (platelet count <150x109 per mL).
* Patients taking long-term Histone Deacetylase Inhibitors such as sodium valproate.
* Patients taking any of the following medications: antipsychotics, MAO inhibitors, antidepressants and benzodiazepines, Lithium, Olanzepine, Phenobarbital, Primidone, Phenytoin, Carbamazepine, Lamotrigine, Felbamate.
* Patients diagnosed with a mitochondrial deficiency disorder.
* Patients with porphyria.
* Patients with known urea cycle disorders.
* Women of child bearing potential (WOCBP) are excluded from the study. A woman is defined as being of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal, unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Patients who are participating in another interventional clinical trial.
* Unable, in the opinion of the investigator, or unwilling to give informed consent protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2024-10-07 (Estimated); Study Completion 2024-10-07 (Estimated)

PRIMARY OUTCOMES:
Change of Serum Creatinine level | Baseline, 2 weeks, 4 weeks, 0-6, 6-12, 24, 48, 72, and 96 hours post-operatively
  Measurement of serum creatinine level and expressed as umol/L.
Change of Serum Troponin I level | Baseline, at 0-6, 6-12, 24, 48 and 72 hours post-operatively
  Measurement of serum Troponin level and expressed as ng/L.

SECONDARY OUTCOMES:
Change in Multiple organ dysfunction - Sepsis-related Organ Failure Assessment (SOFA) Score) | Baseline, 4 weeks, 0-6, 24, 48, 72 and 96 hours
  Range 0-3, 3 being the worse score
NGAL (Neutrophil gelatinase associated lipocalcin) | Baseline, day before surgery, 6-12, 24 and 48 hours post-surgery.
  Measurement of NGAL level and expressed as μg/L.
Lung Injury - Arterial alveolar oxygen (PaO2/FiO2) ratios | Baseline, day before surgery, 24, 48, 72 and 96 hours post-surgery.
  Measurement of PaO2/FiO2 ratio and expressed in kPa/L.
AST (Aspartate Transaminase) | Baseline, day before surgery, 0-6, 6-12, 24, 48, 72 and 96 hours post-surgery
  Measurement of AST levels in serum and expressed in IU/L. Acute liver injury will be defined as an acute derangement of three times the upper limit of normal.
ALT (Alanine Transaminase) | Baseline, day before surgery, 0-6, 6-12, 24, 48, 72 and 96 hours post-surgery
  Measurement of ALT levels in serum and expressed in IU/L. Acute liver injury will be defined as an acute derangement of three times the upper limit of normal.
Bilirubin | Baseline, day before surgery, 0-6, 6-12, 24, 48, 72 and 96 hours post-surgery
  Measurement of Bilirubin levels in serum and expressed in μmol/L. Acute liver injury will be defined as an acute derangement of three times the upper limit of normal.
Alkaline Phosphatase | Baseline, day before surgery, 0-6, 6-12, 24, 48, 72 and 96 hours post-surgery
  Measurement of Alkaline Phosphatase levels in serum and expressed in IU/L. Acute liver injury will be defined as an acute derangement of three times the upper limit of normal.
Serum Amylase | Baseline, day before surgery, 0-6, 6-12, 24, 48, 72 and 96 hours post-surgery
  Measurement of Amylase levels in serum and expressed in IU/L. Acute pancreatitis will be defined as a serum amylase concentration >1000 ng/ml.
Assessment of resource use - Time until extubation | Time (hours) measured from the start of surgery - to extubation (up to 30 days)
Length of stay in Intensive Care Unit | Time (hours) measured from the start of surgery to discharge from ICU (up to 30 days)
  Number of hours between admission and discharge from the Intensive Care Unit (ICU).
Length of Stay in Hospital | Time (days) measured from the start of surgery to discharge from hospital (up to 90 days)
  Number of days between the date of surgery and discharge from the hospital.
Sepsis | Baseline, 4 weeks before surgery, 0-6, 6-12, 24, 48, 72 and 96 hours post-surgery
  Sepsis is defined as: Suspected or documented infection and an acute change in total Sepsis-related Organ Failure Assessment (SOFA) score ≥2 points consequent to the infection. Range of SOFA is 0 to 3, 3 being the worse score.
Rate of mortality | Within 30-days from surgery and at 1 year from surgery
  Rate of mortality at 30-day and 1 year from the date of surgery.
Bleeding and Transfusion | Intra-operative and between time of surgery and hospital discharge up to two weeks
  The total number of units of red cells and other blood components transfused during the operative period and post-operative hospital stay
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Post-operative up to 3 months follow-up from time of surgery
  Adverse events as assessed for type and severity by CTCAE v4.0
Mechanism study: Mithocondrial function of microvessels from tissue biopsies | At time of surgery
  50-100 mg biopsies obtained from pedicled left internal mammary artery biopsies. The mitochondrial function will be measured through the Bioenergetic Health Index. The Bioenergetic Health Index (BHI) is calculated using the following formula: BHI=(ATP-linked×reserve capacity)/(proton leak×non-mitochondrial) - as described by Chacko et al. The expected range is 0-100.
Mechanism study: microRNAs isolation from microvessels | At time of surgery
  The findings will be represented by the frequency (%) of identified microRNAs. 50-100 mg biopsies obtained from pedicled left internal mammary artery biopsies.
Mechanism study: Chromatin Immunoprecipitation (ChIP) of microvessels from tissue biopsies | At time of surgery
  To identify protein binding sites that may help identify functional elements in the genome.
  Findings will be represented by the number (n) of binding sites. 50-100 mg biopsies obtained from pedicled left internal mammary artery biopsies.
Mechanism study: Mithocondrial function measured in right atrium myocardium tissue biopsies | At time of surgery
  50-100 mg myocardial biopsies will be obtained from the right atrium at surgery. The mitochondrial function will be measured through the Bioenergetic Health Index. The Bioenergetic Health Index (BHI) is calculated using the following formula: BHI=(ATP-linked×reserve capacity)/(proton leak×non-mitochondrial) - as described by Chacko et al. The expected range is 0-100.
Mechanism study: microRNA isolation from right atrium myocardium tissue biopsies | At time of surgery
  50-100 mg myocardial biopsies will be obtained from the right atrium at surgery. The findings will be represented by the frequency (%) of identified microRNAs.
Mechanism study: Chromatin Immunoprecipitation (ChIP) in right atrium myocardium tissue biopsies | At time of surgery
  50-100 mg myocardial biopsies will be obtained from the right atrium at surgery. To identify protein binding sites that may help identify functional elements in the genome.
  Findings will be represented by the number (n) of binding sites.
Mechanism study: Mithocondrial function measured in adipose tissue biopsies | At time of surgery
  Adipose tissue collected from epicardial fat at time of surgery. The mitochondrial function will be measured through the Bioenergetic Health Index. The Bioenergetic Health Index (BHI) is calculated using the following formula: BHI=(ATP-linked×reserve capacity)/(proton leak×non-mitochondrial) - as described by Chacko et al. The expected range is 0-100.
Mechanism study: microRNA isolation in adipose tissue biopsies | At time of surgery
  Adipose tissue collected from epicardial fat at time of surgery. The findings will be represented by the frequency (%) of identified microRNAs.
Mechanism study: Chromatin Immunoprecipitation (ChIP) in adipose tissue biopsies | At time of surgery
  Adipose tissue collected from epicardial fat at time of surgery. To identify protein binding sites that may help identify functional elements in the genome.
  Findings will be represented by the number (n) of binding sites.
Mechanism study: Measurement of microvesicles in urine samples | 1 day before surgery, 12 and 24 hours following surgery
  Identification of microvesicles. The findings will be represented by the frequency (%) of each identified microvesicle.
Mechanism study: Measurement of microRNAs in urine samples | 1 day before surgery, 12 and 24 hours following surgery
  The findings will be represented by the frequency (%) of identified microRNAs.
Mechanism study: Measurement of histone acetylation in urine samples | 1 day before surgery, 12 and 24 hours following surgery
  The findings will be reported as acetylated H3 (ug/mg) over time (hours)
Mechanism study: Measurement of gene expression in urine samples | 1 day before surgery, 12 and 24 hours following surgery
  Whole genome sequencing will be achieved through ATAC sequencing. The identified genes will be characterised by average expression count over ATAC.
Mechanism study: Cardiac Magnetic Resonance Imaging - Cardiac Function | Baseline, 1 day before surgery and 3 months following surgery
  Assessment of cardiac function, by assessing ventricular function. This will be expressed as ejection fraction (%). Intravenous contrast will be administered via an indwelling venous catheter.
Mechanism study: Cardiac Magnetic Resonance Imaging - Cardiac adiposity content | Baseline, 1 day before surgery and 3 months following surgery
  Assessment of cardiac adiposity content. A percentage of adipose tissue over total body mass will be calculated. Intravenous contrast will be administered via an indwelling venous catheter.
Mechanism study: Cardiac Magnetic Resonance Imaging - Visceral adiposity content | Baseline, 1 day before surgery and 3 months following surgery
  Assessment of visceral adiposity content. A percentage of adipose tissue over total body mass will be calculated. Intravenous contrast will be administered via an indwelling venous catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Murphy, MD, Study Chair — BHF Professor of Cardiac Surgery, University of Leicester; Marius Roman, MD, Principal Investigator — Academic Clinical Lecturer in Cardiac Surgery, University of Leicester
Locations (1):
- Glenfield Hospital, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No